CLINICAL TRIAL: NCT04433949
Title: Radiation Eliminates Storming Cytokines and Unchecked Edema as a 1-Day Treatment for COVID-19 (RESCUE 1-19): A Randomized Phase III Trial of Best Supportive Care Plus Provider's Choice of Pharmaceutical Treatment With or Without Whole Lung Low-Dose Radiation Therapy (LD-RT) in Hospitalized Patients With COVID-19
Brief Title: Best Supportive Care With or Without Low Dose Whole Lung Radiation Therapy for the Treatment of COVID-19
Acronym: RESCUE1-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mohammad K. Khan, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000781; NCI-2020-04061 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD5049-20 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Pneumonia; Severe Acute Respiratory Syndrome; Symptomatic COVID-19 Infection Laboratory-Confirmed
Keywords: Radiotherapy; COVID-19; low dose radiotherapy; anti-inflammatory; cytokine storm
MeSH Terms: conditions — Pneumonia; Severe Acute Respiratory Syndrome; COVID-19; Cytokine Release Syndrome | interventions — Practice Guidelines as Topic; Standard of Care; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (physician choice) (Active Comparator): Patients get best supportive care + physician choice of treatment
  Interventions: Other: Best Practice
- Arm II (LDRT) (Experimental): Patients receive best supportive care + low dose RT (whole lung)
  Interventions: Radiation: Low Dose Radiation Therapy

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm I (physician choice)
Radiation: Low Dose Radiation Therapy — Undergo LDRT
  Other Names: Low Dose Radiation
  Arms: Arm II (LDRT)

SUMMARY:
This phase III trial compares low dose whole lung radiation therapy to best supportive care plus physicians choice in treating patients with COVID-19 infection. Low dose whole lung radiation therapy may work better than the current best supportive care and physician's choice in improving patients' clinical status, the radiographic appearance of their lungs, or their laboratory blood tests.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Intubation-free survival (IFS) and (2) time to clinical recovery (TTCR) based on weaning off supplementary oxygenation or hospital discharge in COVID 19 patients.

SECONDARY OBJECTIVES:

I. To investigate (1) other clinical, (2) radiographic, (3) serologic markers, and (4) immune marker response to best supportive care plus provider's choice of pharmaceutical treatment either with or without whole-lung LD-RT

II. Secondary clinical improvements will look at time to hospital discharge, prevention of ICU admissions, and overall survival.

OUTLINE: Patients are blindly randomized to 1 of 2 arms.

ARM I: Patients receive best supportive care plus physician choice of treatment

ARM II: Patients receive best supportive care plus LDRT (experimental arm).

After completion of study, patients are followed up for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Be age 50 or over; Not pregnant (will undergo pregnancy testing if below age 55);
* Have had a positive PCR-based test confirming the diagnosis of COVID-19 within 5 days (+/-2 day)of study enrollment*
* Have had clinical signs of severe acute respiratory syndrome or pneumonia (ie. dyspnea, cough,fever) that primary team feels like patient needs rescuing with LD-RT.**
* Have visible bilateral consolidations/ground glass opacities on chest imaging
* Require supplemental oxygen at the time of enrollment, defined by inability to wean from supplemental oxygen within 24 hours prior to enrollment.
* Not require intubation within 12 hours of randomization (ie, not screen fail). Intubation after enrollment but within 12 hours of randomization will be defined as a screen failure for both the LD-RT and control cohorts.
* Be enrolled within 5 days (+/- 2) of first hospitalization for COVID-19. Prior hospitalization for COVID-19 will be an exclusion criteria (prior ED visits are permissible).
* Willingness and ability of the subject to comply with scheduled visits, protocol-specified laboratory tests, other study procedures, and study restrictions
* Evidence of a signed informed consent/assent indicating that the subject is aware of the infectious nature of the disease and has been informed of the procedures to be followed, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation

Exclusion Criteria:

* Pregnant and/or planned to be pregnant within in next 6 months
* Age 49 or younger at time of enrollment
* Prior inpatient hospitalization for COVID-19 (prior emergency department [ED] visits are not an exclusion criteria)
* Prior enrollment on a separate COVID-19-related therapeutric trial (subsequent co-enrollment is permitted for patinets randomized to the control arm).
* Notably, concurrent use of COVID-directed therapies is no longer an exclusion criteria for this trial. This includes azithromycin, dexamethasone, remdesevir, convalescent plasma, or any other COVIDdirected drug therapy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Time to clinical recovery | Up to follow-up day 14 after study start
  Will be measured by improvements on oxygenation need prior to intervention compared with after intervention and/or hospital discharge.

SECONDARY OUTCOMES:
Freedom from ICU admission | Up to follow-up day 14 after study start; This may be extended up to 28 days after preplanned interim analysis.
  The rates from both cohort will be reported.
Temperature | Up to follow-up day 14 after study start
  Temperature in degrees (F)
Heart rate | Up to follow-up day 14 after study start
  Heart rate in beats per minutes
Systolic Blood pressure | Up to follow-up day 14 after study start
  Systolic blood pressure in mm Hg
Oxygen saturation | Up to follow-up day 14 after study start
  Oxygen saturation in percentage
Supplemental oxygenation need | Up to follow-up day 14 after study start
  Oxygen saturation in percentage
Respiratory rate | Up to follow-up day 14 after study start
  Respiratory rate in breaths per minute.
Glasgow Comma Scale from minimum of 3 to maximum of 15. | Up to follow-up day 14 after study start
  Pre and post intervention; Minimum of 3 (poor) to best (15)
Performance status | Up to follow-up day 14 after study start
  Easter Cooperative Oncology Group (ECOG) Performance Status Scale from 0-5; 0 being best; 5 being dead;
Survival | Up to follow-up day 14 after study start; This may be extended to 28 days after preplanned interim analysis.
  Survival in percentage
Serial chest x-rays severe acute respiratory syndrome (SARS) scoring | Up to follow-up day 14 after study start;
  Serial chest x-rays categorized using published scale into ordinal ranks 1-5 for SARS.
Changes on computed tomography (CT) scans pre and post RT | Baseline up to follow-up day 14 after study start
  CT scans with volume of consolidation measured in cubic centimeters.
CRP | Up to follow-up day 14 after study start
  C-Reactive Protein in mg/L
Serum chemistry + complete blood cell (CBC) with differential | Up to follow-up day 14 after study start
  Will be summarized descriptively.
Blood gases pH(when available) | Up to follow-up day 14 after study start
  pH (no unit)
Albumin | Up to follow-up day 14 after study start
  Albumin in gm/dL
Procalcitonin | Up to follow-up day 14 after study start
  Procalcitonin in ng/mL
Aspartate aminotransferase (AST) | Up to follow-up day 14 after study start
  Asparatate Aminotransferase in units/L
Creatine kinase | Up to follow-up day 14 after study start
  Creatinine in mg/dL
Prothrombin time (PT)/partial thromboplastin time (PTT) | Up to follow-up day 14 after study start
  Coagulation pathway time in seconds
Troponin | Up to follow-up day 14 after study start
  Troponin-I in ng/mL
Lactate | Up to follow-up day 14 after study start
  Lactic Acid in mmol/L
NT-pBNP (cardiac injury) | Up to follow-up day 14 after study start
  B-Natriuretic Peptid in pg/mL
Gamma-glutamyl transferase (GGT) | Up to follow-up day 14 after study start
  Gamma-glutamyl transferase in units/L
Triglycerides | Up to follow-up day 14 after study start
  Trygliciericdes in mg/dL
Fibrinogen | Up to follow-up day 14 after study start
  Fibrinogen in mg/dL
Changes in CD8 T cells | Up to follow-up day 14 after study start
  Will be summarized descriptively.
Changes in CD4 T cells | Up to follow-up day 14 after study start
  Will be summarized descriptively.
Changes in serum antibodies against COVID-19 epitope | Up to follow-up day 14 after study start
  Will be summarized descriptively.
LDH | Up to follow-up day 14 after study start
  Lactate Dehydrogenase in units/L
D-Dimer | Up to follow-up day 14 after study start
  D-Dimer in ng/mL
IL-6 | Up to follow-up day 14 after study start
  Interleukin-6 in pg/mL
Myoglobin | Up to follow-up day 14 after study start
  Myoglobin in ng/mL
Potassium | Up to follow-up day 14 after study start
  Potassium in mmol/L
Ferritin | Up to follow-up day 14 after study start
  Ferritin in ng/mL
ALT | Up to follow-up day 14 after study start
  Alanine Aminotransferase in units/L

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad K Khan, MD, PhD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Results of the trial and not individual patient data will be shared. The study protocol, consent, and investigator's brochure will be available. The statistical plan is incorporated into the protocol, along with inclusion and exclusion criteria.

REFERENCES:
- [Background] Lara PC, Burgos J, Macias D. Low dose lung radiotherapy for COVID-19 pneumonia. The rationale for a cost-effective anti-inflammatory treatment. Clin Transl Radiat Oncol. 2020 Apr 25;23:27-29. doi: 10.1016/j.ctro.2020.04.006. eCollection 2020 Jul. PMID 32373721
- [Background] Dhawan G, Kapoor R, Dhawan R, Singh R, Monga B, Giordano J, Calabrese EJ. Low dose radiation therapy as a potential life saving treatment for COVID-19-induced acute respiratory distress syndrome (ARDS). Radiother Oncol. 2020 Jun;147:212-216. doi: 10.1016/j.radonc.2020.05.002. Epub 2020 May 8. PMID 32437820
- See also: Interim Results from the phase 1, 2 pilot safety trial of LD-RT for COVID — https://www.medrxiv.org/content/10.1101/2020.06.03.20116988v1
- See also: Article on Forbes — https://www.forbes.com/sites/jamesconca/2020/06/12/1st-human-trial-successfully-treated-covid-19-using-low-doses-of-radiation/#34a56312dc69